CLINICAL TRIAL: NCT02607657
Title: Phase I Trial Comparing Eplerenone Pharmacokinetics (Tablet) in Different Dosages: 25mg, 50mg,100 mg Per Day and 100 mg (One 50 mg Tablet Every 12 Hours).
Brief Title: Pharmacokinetics of Eplerenone Tablet
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GDN 055/15
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Eplerenone 25 mg (Experimental): Eplerenone 25 mg Tablet Oral Once daily
  Interventions: Drug: Eplerenone 25 mg
- Eplerenone 50 mg (Experimental): Eplerenone 50 mg Tablet Oral Once daily
  Interventions: Drug: Eplerenone 50 mg
- Eplerenone 100 mg (Experimental): Eplerenone 100 mg (2 tablets of 50 mg) Tablet Oral Once daily
  Interventions: Drug: Eplerenone 100 mg
- Eplerenone 50 mg x 2 (Experimental): Eplerenone 50 mg Tablet Oral Twice daily
  Interventions: Drug: Eplerenone 50 mg twice a day
- Eplerenone 25 mg x 2 (Experimental): Eplerenone 25 mg Tablet Oral Twice daily
  Interventions: Drug: Eplerenone 25 mg twice a day

INTERVENTIONS:
Drug: Eplerenone 25 mg
  Arms: Eplerenone 25 mg
Drug: Eplerenone 50 mg
  Arms: Eplerenone 50 mg
Drug: Eplerenone 100 mg
  Arms: Eplerenone 100 mg
Drug: Eplerenone 50 mg twice a day
  Arms: Eplerenone 50 mg x 2
Drug: Eplerenone 25 mg twice a day
  Arms: Eplerenone 25 mg x 2

SUMMARY:
This is a Phase I, open-label, randomized, parallel trial to evaluate the pharmacokinetics of Eplerenone tablet at different dosages (25 mg once daily, 50 mg once daily, 100 mg (2 tablets of 50 mg) once daily and 50 mg twice daily). Sample size is 96 participants (24 per treatment group), male or female, aged between 18 and 50 years-old.

Primary objective is to evaluate pharmacokinetics of Eplerenone tablet at different dosages, and secondary objective is to evaluate safety and tolerability of the investigational product.

Study overall duration is approximately 12 weeks, including enrollment and follow-up visits. Participants will be admitted for a period of 36 hours, when investigational product will be administered, and blood samples, at pre-determined time periods, will be collected for pharmacokinetics.

Primary endpoint is to obtain pharmacokinetics parameters. Additionally, safety will be assessed by adverse events occurrence and laboratory exams evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female study participants, aged between 18 and 50 years-old;
* Healthiness, according to clinical, laboratory and electrocardiographic evaluations;
* Ability to understand the nature and objectives of the trial, including risks and adverse events; willingness to cooperate with the researcher and proceed according to all study requirements, which shall be confirmed by Informed Consent Form signature.

Exclusion Criteria:

* Known hypersensitivity to the investigational product (Eplerenone) or chemically related compounds; history of serious adverse reactions or hypersensitivity to any drug;
* History or presence of hepatic or gastrointestinal diseases, or other condition that interferes with drug absorption, distribution, excretion or metabolism;
* Chronic therapy with any drugs, except oral contraceptives;
* History of hepatic, kidney, lungs, gastrointestinal, epileptic, hematologic or psychiatric disease; hypotension or hypertension, of any etiology, that requires pharmacological treatment; history of myocardial infarction, angina and/or heart failure;
* Electrocardiographic findings that, at investigator criteria, are not recommended for study participation;
* Deviations on screening laboratory results that are considered clinically relevant by the researcher, preventing the subject to participate in the trial;
* Smoking;
* Intake of more that 5 cups of coffee or tea per day;
* Unusual food habits, e.g., vegetarians;
* History of drugs and alcohol addiction or excessive alcohol consumption (> 35 g/day);
* Use of regular medications within 2 weeks prior study enrollment or use of any medications within one week prior to study enrollment, except oral contraceptives or cases which, based on drug's or metabolite's half-life, complete elimination can be assumed;
* Hospitalization for any reasons up to 8 weeks before trial;
* Treatment, within 6 months before the trial, with any drugs with known and well-established toxic potential to major organs;
* Participation in any other experimental research or administration of any experimental drug within 3 months before this trial;
* Donation or loss of 450 mL or more of blood within 3 months before this trial or 3 donations (women)/4 donations (men) of blood within 12 months before this trial;
* Any condition, according to investigator's best judgement, that prevents the subject to participate in the trial;
* Pregnancy, labor or miscarriage with 12 weeks before admission predicted date.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Area under the curve(0-last) | 24 hours
Area under the curve(0-all) | 24 hours
Area under the curve(0-inf) | 24 hours
Half-life (t1/2) | 24 hours
Elimination rate constant (Ke) | 24 hours
Maximum serum concentration (Cmax) | 24 hours
Time to reach maximum (peak) plasma concentration following drug administration (tmax) | 24 hours
Time of the last measurable (positive) concentration (tlast) | 24 hours
Area under the first moment of the plasma concentration-time curve extrapolated from time zero to infinity as a percentage of total AUC | 24 hours

SECONDARY OUTCOMES:
Number of adverse events | 30 days
Intensity of adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, PhD, Principal Investigator — Galeno Desenvolvimento de Pesquisas Ltda.